CLINICAL TRIAL: NCT00618124
Title: A Phase 1 Safety And Pharmacokinetic Study Of SU011248 And Capecitabine In Patients With Advanced Solid Tumors
Brief Title: A Study To Find The Best Doses Of SU011248 (Sunitinib) And Capecitabine When These Drugs Are Administered Together
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181044
Record Dates: First submitted 2008-02-01; First posted 2008-02-18 (Estimated); Last update posted 2010-05-03 (Estimated); Status verified 2010-04

CONDITIONS: Solid Tumors; Breast Cancer; Neoplasms
Keywords: solid tumor malignancy, SU011248, sunitinib, capecitabine, Phase 1
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Sunitinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: SU011248; Capecitabine

INTERVENTIONS:
Drug: SU011248; Capecitabine — Dose finding study using SU011248 daily by oral capsule in a continuous regimen or administered for 4 out of every 6 weeks (Schedule 4/2) or 2 out of every 3 weeks (Schedule 2/1), with capecitabine administered 2 out of every 3 weeks until progression or unacceptable toxicity.
  Other Names: Sutent, sunitinib, SU11248, Xeloda

SUMMARY:
This study assesses the maximum tolerated dose, overall safety and antitumor activity of SU011248 in combination with capecitabine in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of a solid cancer which is not responsive to standard therapy or for which no standard therapy exists
* Patient has good performance status (ECOG 0 or 1)

Exclusion Criteria:

* Prior treatment with either SU011248 or capecitabine.
* Hypertension that cannot be controlled by medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximally tolerated dose of SU011248 (dosed continuously or on a 4/2 or 2/1 Schedule) when given in combination with capecitabine. | From Screening until disease progression or discontinuation of the study

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of SU011248 and capecitabine when these drugs are co-administered | From Cycle 1, Day 1 until discontinuation of the study
To preliminarily assess the antitumor activity of SU011248 and capecitabine in patients with measurable disease | From screening until disease progression or discontinuation of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Albuqurque, New Mexico
  - Pfizer Investigational Site, Nashville, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181044&StudyName=A%20Study%20To%20Find%20The%20Best%20Doses%20Of%20SU011248%20%28Sunitinib%29%20And%20Capecitabine%20When%20These%20Drugs%20Are%20Administered%20Together